CLINICAL TRIAL: NCT03995745
Title: Behavioral Economic Incentives to Improve Medication Adherence and Outcomes Among Patients in United States With HIV: A Feasibility Study
Brief Title: Medication Adherence and Outcomes Among Patients in United States With HIV
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 831689
Record Dates: First submitted 2019-05-23; First posted 2019-06-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Human Immunodeficiency Virus; Medication Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Intervention Model Description: HIV-positive patients in Philadelphia with non-suppressed viral loads will be randomly assigned to receive the intervention (electronic-pill bottle with adherence based daily financial incentives, and incentive for reaching viral suppression) or control. About 40 patients will be enrolled in the study, 20 in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adherence based financial incentives (Experimental): Participants randomized to this arm will receive an electronic pill bottle, AdhereTech. The AdhereTech bottle will be remotely monitored by the Way to Health platform. Participants will be randomly assigned a 2-digit number to be used as part of the lottery-based engagement incentives in which eligibility to win will be conditional on medication adherence. Participants will also be eligible for a financial bonus if participant's viral load is suppressed at the end of the intervention period. Participants will also receive an enrollment incentive and an incentive to complete a lab visit at the end of the intervention period.
  Interventions: Behavioral: Medication adherence and financial incentives
- control (No Intervention): Of the 20 participants randomized to the control arm, 10 will be randomly assigned to receive an electronic pill bottle, AdhereTech. The AdhereTech bottle will be remotely monitored by the Way to Health platform. Participants will also receive an enrollment incentive and an incentive to complete a lab visit at the end of the intervention period.

INTERVENTIONS:
Behavioral: Medication adherence and financial incentives — Provision of wireless devices and financial incentives to motivate medication adherence among HIV-positive adults who have not reached viral suppression.
  Arms: adherence based financial incentives

SUMMARY:
With support from the NIH, this pilot study will assess the feasibility of using wireless devices and financial incentives to motivate medication adherence among HIV-positive adults in the U.S., focusing on those with non-suppressed viral loads.

While daily lotteries using wireless devices may have great potential for improving adherence to ART regimens, substantial questions exist as to whether it is: 1) possible to achieve high rates of uptake for a pilot offering wireless devices to high-risk populations; 2) achieve high rates of sustained engagement.

DETAILED DESCRIPTION:
The goal of this study is to explore the feasibility of using wireless devices and financial incentives to motivate medication adherence among high-risk HIV positive patients. By partnering with the Drexel Partnership Comprehensive Care Clinic at Drexel University, the investigators will be able to identify such patients using clinic patient data, use clinic and physician communication channels to enroll them, and maintain high levels of ongoing participation through the use of incentives. The aim is to improve antiretroviral medication adherence among high-risk HIV positive patients by providing patients with a AdhereTech device (electronic pill bottle), daily adherence notifications tracked by the Way to Health platform, as well as daily lotteries and financial incentives. Upon completion, this study will answer questions important to the feasibility of conducting well-powered randomized controlled trials to improve adherence among HIV patients within the U.S. who have sub-optimal adherence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV, established in 2017 or earlier
* Patients at least 18 years of age or older
* Currently prescribed first or second line ART medications
* Non-suppressed viral loads, with two consecutive non-suppressed viral loads (VL>400 copies/ml) for the past two lab readings.

Exclusion Criteria:

* Pregnant
* Prescribed Maraviroc or Fuzeon
* More than 5 additional medications
* Diagnosed with insulin dependent diabetes
* Unable to provide consent
* Non-English speaker
* Cognitive impairment, per PI discretion
* Does not have stable residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with viral suppression | approximately 3 months after enrollment
  viral load less than 400

SECONDARY OUTCOMES:
viral suppression by arm | approximately 3 months after enrollment
  viral load less than 400
medication adherence by arm | approximately 3 months after enrollment
  electronic pill bottle openings by day
Recruitment rates by arm | approximately 3 months after enrollment
Attrition rates by arm | approximately 3 months after enrollment
Percent of patients that use electronic pill bottle | approximately 3 months after enrollment
Completion rates of lab visit by arm | approximately 3 months after enrollment
number of clinic visits by arm | approximately 3 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bien-Gund CH, Ho JI, Bair EF, Marcus N, Choi RJ, Szep Z, Althoff A, Momplaisir FM, Thirumurthy H. Brief Report: Financial Incentives and Real-Time Adherence Monitoring to Promote Daily Adherence to HIV Treatment and Viral Suppression Among People Living With HIV: A Pilot Study. J Acquir Immune Defic Syndr. 2021 May 1;87(1):688-692. doi: 10.1097/QAI.0000000000002628. PMID 33470727